CLINICAL TRIAL: NCT01765647
Title: Use of an Orally Administered Antibody to Gluten to Prevent the Recurrence of Symptoms and Laboratory Parameters in Persons With Celiac Disease (Gluten Sensitive Enteropathy)
Brief Title: Oral AGY for Celiac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Igy Inc. (Industry)
Collaborators: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGY
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-10

CONDITIONS: Celiac Disease
Keywords: Celiac disease; AGY
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: All participants received open label AGY, a natural health product
Oversight: Data Monitoring Committee: No

ARMS (1):
- AGY (Experimental): All participants will receive the same, open-label dose of AGY
  Interventions: Other: AGY

INTERVENTIONS:
Other: AGY — AGY is a natural health product produced in egg yolks

SUMMARY:
Celiac disease (CD) is an autoimmune disease of the small intestine caused by the consumption of gluten proteins from widely used food sources such as wheat, rye, and barley. Exposure of the small intestine to gluten causes an inflammatory response, leading to the destruction of intestine lining, often with severe symptoms including diarrhea, abdominal distention, fatigue, weight loss, anemia, and neurological symptoms. CD is a lifelong disease and the only treatment currently available is strict adherence to a life-time gluten free diet (GFD). However, adhering to this diet is difficult as gluten proteins are found in many food products. Therefore, the gluten-free diet has both lifestyle and financial implications for the individual and thus has been potential for impacting adversely on their quality of life.

Various approaches are being studied to reduce the need for careful control of the diet for those with CD, including the use of antibodies such as IgY. IgY is produced from the egg yolks of super immunized laying hens. Egg yolk antibodies are natural products with minimal toxicity, for those without egg allergy, and offer low-cost, hygienic production of study product. Once the IgY antibody is put into capsule form, it is called AGY.

Individuals with CD will be recruited only if they have a history of biopsy proven CD, currently follow a GFD but continue to have mild to moderate symptoms related to gluten exposure, and do not have an egg allergy. Blood will be tested for ATG antibody levels at screening. Those enrolled will have a 2 week run-in period where diet and symptoms are recorded, and will then receive AGY capsules to take with meals over a 4 week period. Outcomes will be measured by examining lab test results including antibody levels, symptoms, and quality of life.

DETAILED DESCRIPTION:
The trial will last approximately 6 weeks. Individuals will be screened to ensure they are following a gluten free diet, continue to have mild to moderate symptoms of gluten exposure despite the diet, and have a history of biopsy proven celiac disease. Those meeting this criteria will then have a baseline visit which will include a short physical exam and additional lab work for safety measures, and quality of life questionnaires. They will record their diet and symptoms for 2 weeks, and then return to receive the study medication, which will be taken with all meals. The first dose will be taken in clinic to facilitate observation of any adverse effects. The next visit will be 2 weeks later for blood work and clinic visit, and then again 2 weeks later for the final visit. Participants will be prompted to report any adverse events that occur during the trial period and at the completion of the trial. During the trial period, the study coordinator will phone participants to remind them to complete their questionnaires and to inquire about adverse events. All participants will receive AGY capsules (500 mg per capsule), and will take 2 capsules with each meal.

Outcome measures The primary outcome variable will be the safety (adverse events, lab results, symptoms), which will be measured throughout the study.

The secondary outcome will be ATG antibody levels, which will be measured at each visit.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or over
* confirmed diagnosis of Celiac disease by previous biopsy
* follow a gluten-free diet (GFD)
* have mild to moderate symptoms despite the GFD diet

Exclusion Criteria:

* diabetic
* use of steroids in previous year
* current use of ASA/NSAIDs, metronidazole, or misoprostol
* excess alcohol intake
* egg allergy
* history of severe complications of celiac disease or chronic active GI disease
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Dieleman, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- AGY: Anti-gliadin Antibody for Celiac Disease: All participants will receive the same, open-label dose of AGY
  AGY: AGY is a natural health product produced in egg yolks
Period: Overall Study
Arm/Group | AGY: Anti-gliadin Antibody for Celiac Disease
Started | 10 (One began the run-in period, but was withdrawn prior to beginning treatment with AGY)
Completed | 10 (10 entered the AGY treatment phase and all 10 completed treatment.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AGY: Anti-gliadin Antibody for Celiac Disease
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 43.4 [29 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
Region of Enrollment [Number; unit: participants]
  Canada | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Which Treatment Was Concluded to be Safe
Description: Measures include: adverse events, serious adverse events, withdrawal due to adverse events, abnormal lab results
Time Frame: week 6
Measure: Number; unit: participants
Arm/Group | AGY: Anti-gliadin Antibody for Celiac Disease
Number analyzed (Participants) | 10
participants
  mild adverse events during run-in | 6
  moderate adverse events during run-in | 18
  severe adverse events during run-in | 4
  mild adverse events on tx week 2-4 | 5
  moderate adverse events on tx week 2-4 | 11
  severe adverse events on tx week 2-4 | 2
  mild adverse events on tx week 4-6 | 5
  moderate adverse events on tx week 4-6 | 1
  severe adverse events on tx week 4-6 | 3
  serious adverse events at any time | 0
  withdrawal due to adverse event at any time | 0
  all cause mortality | 0

2. Secondary Outcome: Number Celiac Disease Related Symptoms in Participants
Description: Symptoms of Celiac disease will be self-measured by participants daily for the entire 6 week study period using the Celiac Symptom Index tool.
Time Frame: daily for 6 weeks
Measure: Number; unit: Number of Celiac Disease Related Symptom
Arm/Group | AGY: Anti-gliadin Antibody for Celiac Disease
Number analyzed (Participants) | 10
Number of Celiac Disease Related Symptom
  tiredness during 2 weeks of run-in | 93
  tiredness during last 2 weeks on AGY | 52
  headache during 2 weeks of run-in | 59
  headache during last 2 weeks on AGY | 39
  abdominal pain/discomfort during 2 weeks of run-in | 48
  abdominal pain/discomfort during last 2 weeks on A | 39
  bloating during 2 weeks of run-in | 45
  bloating during last 2 weeks on AGY | 26

3. Secondary Outcome: Health Related Quality of Life
Description: health related quality of life will be measured at 4 time points using a validated tool; (short form 36; SF-36) baseline, week 2, week 4, and at the end of the study at week 6.
  Scores can range from 20-80, with 50 being a population norm. Therefore, a score above 50 indicates better than the general population norm, and a score below 50 indicates worse than the population norm.
Time Frame: week 6
Population: Scores were assessed at baseline, week 2, week 4 and week 6; baseline and week 6 reported.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | AGY: Anti-gliadin Antibody for Celiac Disease
Number analyzed (Participants) | 10
score on a scale
  baseline physical component summary | 50.08 [20 to 80]
  week 6 physical component summary | 51.77 [20 to 80]
  baseline mental component summary | 49.34 [20 to 80]
  week 6 mental component summary | 52.12 [20 to 80]

4. Secondary Outcome: ATG Antibody Level
Description: The ATG antibody level will be measured at baseline, week 2, week 4 and week 6. Normal values are less than 7; elevated values mean a worse outcome. Assessed at baseline, week 2, week 4 and week 6; baseline and week 6 reported.
Time Frame: screening through final visit
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | AGY: Anti-gliadin Antibody for Celiac Disease
Number analyzed (Participants) | 10
U/mL
  baseline IgA TTG | 1.538 (1.128)
  week 6 IgA TTG | 0.922 (0.606)

ADVERSE EVENTS:
Arm/Group | AGY: Anti-gliadin Antibody for Celiac Disease
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGY: Anti-gliadin Antibody for Celiac Disease (N=10)
tiredness (General disorders) | 1
abdominal discomfort (Gastrointestinal disorders) | 7
sore ear (Ear and labyrinth disorders) | 1
itchy or red eyes (Eye disorders) | 2
sphincter of oddi syndrome (Hepatobiliary disorders) | 1
cold symptoms (Infections and infestations) | 3
muscle discomfort (Musculoskeletal and connective tissue disorders) | 4
headache (Nervous system disorders) | 6
menstrual cramps (Reproductive system and breast disorders) | 1
conjestion or sore throat (Respiratory, thoracic and mediastinal disorders) | 7
eczema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No